CLINICAL TRIAL: NCT00404716
Title: Effects of Triple Versus Dual Antiplatelet Therapy in Patients With Acute Coronary Syndrome Undergoing Coronary Stent Implantation
Brief Title: Triple Versus Dual Antiplatelet Therapy in Patients Undergoing Coronary Stent Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH-2006-A006
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Cilostazol

INTERVENTIONS:
Drug: Cilostazol

SUMMARY:
Cilostazol is an kind of oral antiplatelet agent with a rapid onset of action that selectively inhibits phosphodiesterase III, a mechanism different from adenosine diphosphate (ADP) receptor antagonists. Previous studies had suggested that cilostazol has lipid-modifying and vasodilating effects in addition to antiplatelet effects. From those experimental and clinical backgrounds, we assumed that triple antiplatelet therapy with aspirin, clopidogrel, and cilostazol might have a beneficial effect on the prevention of atherothrombosis complications following coronary stenting. Therefore, we evaluated the safety and efficacy of triple antiplatelet regimen of aspirin, clopidogrel and cilostazol compared with dual antiplatelet regimen of aspirin and clopidogrel in patients with acute coronary syndrome undergoing successful coronary artery stenting.

Patients undergoing successful coronary stenting were divided into dual antiplatelet therapy (aspirin plus clopidogrel) and triple antiplatelet therapy (aspirin and clopidogrel plus cilostazol) groups. All enrolled patients in triple regimen group will receive cilostazol 100mg, b.i.d., for 6 months in addition to standard dose and duration of aspirin and clopidogrel for post-PCI. The primary endpoints included death, myocardial infarction, target lesion revascularization, stent thrombosis within 30 days, binary restenosis at six month and major adverse cardiac events (MACE) at one year. The secondary endpoints were side effects of study drugs, including major bleeding, vascular complication, hypersensitivebility, and bleeding complications. The study will be powered to test the hypothesis that triple antiplatelet therapy is better than dual antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ACS Undergoing coronary stent implantation
* Between ages of above 18 Years and bellow 80 Years.
* Presence of one or several stenosis in native coronary arteries requiring PCI.
* Willing and able to sign informed consent.

Exclusion Criteria:

* A history of bleeding diathesis.
* New York Heart Association functional class IV.
* Prior PCI or coronary bypass grafting < 3 months.
* Contraindications to clopidogrel and aspirin (White blood cells counts < 4×109/L or platelet counts <100 g.l-1 ;creatinine clearance <25 ml • min-1 ;active liver disease).
* Use of glycoprotein IIb/IIIa inhibitors before PCI.
* Preparing to undergo CABG
* Taken clopidogrel or cilostazol recently

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Dr., Principal Investigator — Shenyang Northern Hospital